CLINICAL TRIAL: NCT00688272
Title: A Phase I, Double-blind, Placebo and Observer-blind Positive Controlled, Randomized, Parallel Group Study in Healthy Subjects to Investigate the Photoirritant Potential of Eltrombopag
Brief Title: Study In Healthy Subjects To Evaluate The Photo-Irritant Potential Of Eltrombopag
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TRA106914
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: Safety; Photoirritant; Photosensitivity; Placebo control; Ciprofloxacin; Eltrombopag
MeSH Terms: conditions — Purpura; Photosensitivity Disorders | interventions — Ciprofloxacin; eltrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm 1 (Experimental): Eltrombopag 75 mg QD x 6 days
  Interventions: Drug: Eltrombopag
- Arm 2 (Active Comparator): Ciprofloxicin 500mg BID x 6 days
  Interventions: Drug: Ciprofloxacin
- Arm 3 (Placebo Comparator): Placebo QD x 6 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — Given 500mg BID x 6 days
  Arms: Arm 2
Drug: Eltrombopag — Given QD x 6 days
  Other Names: Ciprofloxacin
  Arms: Arm 1
Drug: Placebo — Given QD x 6 days
  Arms: Arm 3

SUMMARY:
This study is designed to investigate the safety profile and the photoirritant potential of eltrombopag in healthy subjects. The study is placebo- and positive controlled, randomized, parallel group with three treatment arms: eltrombopag (75 mg QD), placebo, and a positive control (ciprofloxacin, 500 mg BID). Eltrombopag will be administered in a double-blind fashion with respect to placebo and the positive control, ciprofloxacin, will be administered under observer-blinded conditions. Twelve to fifteen subjects will be recruited into each arm, to assure total enrollment of 36 evaluable subjects. The primary endpoint is the photosensitizing potential of eltrombopag as measured by photoirritant index (PI) and change in minimum erythemal dose (MED) in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male or females with no clinically significant abnormality identified by the physician by evaluation of medical history, physical examination, clinical laboratory tests or 12-lead ECG.
* Subjects were adult males or females between 18 and 65 years of age, inclusive.
* All female subjects of child bearing potential agreed to commit to one of the protocol approved methods of contraception, and that they were used consistently and in accordance with both the product label and the instructions of a physician. Female participants are not permitted to use Hormonal form of contraception (combined oral contraceptive pills etc) because of its known potential to induce photosensitivity.
* All male subjects agreed to abstain completely from (or use a condom during) sexual intercourse with a pregnant or lactating female.
* All male subjects with partner(s) who is /are able to have children agreed to use condom with spermicide from screening until 90 days after the last dose of study medication. In addition, their partner (s) had to also use one of the following forms of contraception until 90 days after last date of study medication:
* Hormonal contraception i.e. the pill or hormones given by injection or given under the skin.
* Diaphragm with spermicide
* Cervical cap or female condoms.
* An intrauterine device (a coil micro-insert).
* Intrauterine system (IUS) e-g Mirena coil
* Tubal ligation
* Body weight greater than or equal to 50 kg and body mass index within the range 19-29.9 kg/m2.
* A signed and dated written informed consent was obtained for the subject.
* Skin Type 1, 2, or 3 according to the dermatological scale presented in the study protocol (see Modular Appendices).
* Negative test for porphyrins, ANF, anti-Ro and anti-La (tests for lupus erythematosus) at screening.
* Liver function tests (LFTs; AST, ALT, ALP, bilirubin, gamma-GT) within the reference range, or deviations that were not considered clinically significant at screening by the investigator.
* Subjects who had a normal value of MED in comparison with the normal population databank at the photobiology unit, Dundee.
* The subject was able to understand and comply with protocol requirements and time tables, instructions and protocol-stated restrictions Exclusion Criteria
* Any abnormality identified on the screening medical assessment that in the opinion of the investigator and GlaxoSmithKline medical monitor could have been associated with an increased rish to the subject or could have interfered with study procedures.
* Subjects who had any sun or sunbed exposure to the skin of the back during the four weeks prior to the screening period.
* Subjects with history of polymorphic light eruption.
* Subjects who had a history of sensitivity to ciprofloxacin, any of the study medications or components thereof.
* Subjects with history of malignant melanoma in a first degree family member.
* Subjects with history of Gilbert Syndrome.
* Subjects with history of deep vein thrombosis or any other thromboembolic event.
* Subjects with history of sensitivity to heparin, or heparin-induced thrombocytopenia.
* Subjects with history of platelet clumping that prevents reliable measurement of platelet counts.
* Subjects with history of thrombocytopenia or bleeding due to abnormal platelet number or function.
* Subjects with C-reactive protein (CRP) that is elevated above normal range and considered clinically significant at screening.
* Subjects with history of myocardial infarction, stroke or sudden unexplained death in a first degree family member under the age of 60 years.
* Subjects with clotting factor abnormalities associated with hypercoagulability, specifically Factor V Leiden, Protein C, or Protein S deficiency, or antithrombin III deficiency.
* Subjects with haemoglobin, white blood cells, platelet count or reticulocyte count that are outside the reference range and considered clinically significant at screening by the investigator.
* Subjects with positive test for HIV, hepatitis B virus or hepatitis C virus.
* Subjects with positive urine drug screen including alcohol.
* Subjects with history of alcohol/drug abuse or dependence within 12 months of screening.
* History of regular alcohol consumption exceeding average weekly intake of greater than 21 units or an average daily intake of greater than three units (males) or an average weekly intake of greater than 14 units or an average daily intake of greater than two units (females). One unit is equivalent to a half-pint (220 mL) of beer/lager or one (25 mL) measure of spirits or one glass (125 mL) of wine.
* Subjects who could not refrain from smoking during the study period from Day-1 through the completion of follow-up assessments.
* Subjects who had received treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
* Subjects who had been exposed to more than four new chemical entities within 12 months prior to the first dosing day.
* Subjects who had taken any prescription or non-prescription drugs (including aspirin and NSAIDs), vitamins, herbal and dietary supplements, or any herbal remedies containing St. John's Wort within seven days (or 14 days if the drug is a potential enzyme inducer) or five half-lives (whichever is longer) prior to the first dose of study medication and through the completion of follow-up assessments. By exception, acetaminophen (or, paracetamol) at doses of less than or equal to 2 g/day and stable thyroid replacement therapy was allowed.
* Consumption of antacids (e.g., Maalox, Mylanta, Amphogel, Milk of Magnesia or TUMS™) within 48 h of the first dose of study medication and until the completion of follow-up assessments.
* Subjects who had an clinically significant skin/allergic disease, including photo-allergy (excluding non

  * active hay fever).
* Subjects with multiple tattoos which may have obscured skin reactions or which restricted the skin surface area available for testing.
* Subjects had to abstain from consumption of grapefruit, pomelo or Seville oranges from screening until the completion of follow-up assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-06-02 (Actual); Primary Completion 2008-09-25 (Actual); Study Completion 2008-09-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the photosensitizing potential, as measured by photoirritant index and change from baseline in minimum erythemal dose, of eltrombopag when dosed orally at 75 mg QD as compared to placebo and ciprofloxacin 500 mg BID. | Screening - Day 8

SECONDARY OUTCOMES:
Severity of phototoxic response Concentration of porphyrins, ANF, anti-Ro, and anti-La as measured on Day 6. | Day 6
Vital signs (blood pressure, heart rate, respiration rate and body temperature) taken after resting semi-supine position for at least 10 minutes; | Screening, Days 1,2,3,4,5,6,7, and f/u
Clinical laboratory tests | Screening, Day 1, 7 and f/u
Assessment of AEs. | Continuous trhoughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dundee, United Kingdom

REFERENCES:
- [Background] Bowen CJ, Lobb KM, Park JW, Sanderson B, Ferguson J. Eltrombopag (75 mg) does not induce photosensitivity: results of a clinical pharmacology trial. Photodermatol Photoimmunol Photomed. 2010 Oct;26(5):243-9. doi: 10.1111/j.1600-0781.2010.00538.x. PMID 20831698
- See also: Results for study TRA106914 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/TRA106914?search=study&search_terms=106914#rs